CLINICAL TRIAL: NCT02499601
Title: CORolla® TAA for Heart Failure With Preserved Ejection Fraction (HFpEF) and Diastolic Dysfunction (DD) Safety and Feasibility
Brief Title: CORolla® TAA for Heart Failure With Preserved Ejection Fraction (HFpEF) and Diastolic Dysfunction (DD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CorAssist Cadiovascular Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD_CRL_0403
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-06

CONDITIONS: Diastolic Heart Failure; Diastolic Dysfunction
Keywords: Heart Failure with Preserved Ejection Fraction (HFpEF); Heart Failure (HF); New York Heart Association functional Class (NYHA f. Cl)
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

ARMS (1):
- CORolla™ TAA Stand Alone (Experimental): Single arm study design including with patients with isolated HFpEF, in NYHA f. Cl. III-IV. These patients will receive the CORolla™ TAA device. For assessments of results, intra-patient comparisons of pre-procedure and follow-up data will be performed;
  Interventions: Device: CORolla™ TAA device

INTERVENTIONS:
Device: CORolla™ TAA device

SUMMARY:
The study objective is to demonstrate safety and feasibility of the CORolla® TAA during 12 months of follow up, and to evaluate the performance of the therapy in relieving symptoms and restore diastolic function in patients with heart failure and preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria

Clinical criteria:

1. Adult (age > 18 years)
2. Diagnosis of heart failure with preserved ejection fraction
3. NYHA F. Class III or IV or documented history of at least two heart failure hospitalization in the past year prior to enrollment.
4. No contraindication for anticoagulation and antiplatelet treatment.
5. Optimal medical cardiovascular pharmacotherapy with stable doses for at least 4 weeks (not including diuretics)
6. Pulmonary Wedge pressure > 15 mmHg documented by right heart catheterization at enrollment.
7. Patient understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
8. Patient is able and willing to adhere to the required follow-up visits and testing
9. Minimal endocardial height from Apex to Mitral Annulus > 60mm at end systole

Echocardiographic criteria:

1. Left ventricular ejection fraction≥50%
2. HFpEF diagnosis according to ESC 2016 guidelines
3. No evidence of intra-cardiac thrombus

Cardiovascular disease:

1. Implanted or planned implantation of defibrillator devices such as ICD cardiac resynchronization device (CRT-D) or left ventricular assist device (LVAD).
2. Within the past 3 months - Acute myocardial infarction (AMI), cerebral vascular accident (CVA), or Transient Ischemic Attack (TIA).
3. History of thrombus within the previous 3 months.
4. Coronary Artery Bypass Surgery (CABG), valve replacement or repair, aortic surgery or percutaneous coronary intervention (PCI in the past 3 months or planned/anticipated within the coming 6 months. Patients with mechanical valve replacement or CABG performed more than 3 months before may be eligible for enrollment.
5. Significant valvular disease classified as

   * Moderate or severe aortic stenosis/regurgitation
   * Moderate or severe mitral stenosis
   * Severe mitral regurgitation
6. Hypertrophic cardiomyopathy
7. History of pericardial disease.
8. HF attributed to Cor pulmonale or other cause of isolated right heart failure.
9. Moderate to severe right ventricle failure or right ventricular myocardial infarction.
10. Infiltrative heart disease including amyloidosis.

Non-cardiovascular disease:

1. Prior surgery, radiation, or thoracic surgery limiting the ability to place the device.
2. Moderate to severe asthma or COPD, or severe restrictive lung disease.
3. Severe chronic renal failure indicated by MDRD GFR <30 mL/min/1.73 m2.
4. Liver impairment addressed by bilirubin > 2 mg/dl and serum albumin <3 g/dL
5. Severe anemia addressed by Hb concentration <9 gr/l.
6. Solid organ or hematologic transplant.
7. Previous Trans Apical procedures/implantation.

Miscellaneous conditions:

1. Co-morbid condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
2. Pregnancy at the time of enrollment. (Women of childbearing potential must have a negative serum pregnancy test within two weeks prior to enrollment, or be using hormonal contraceptives or intrauterine devices).
3. Participating in another treatment investigational study.
4. A history of alcohol abuse, drug addiction, or other psychosocial condition that would preclude successful participation, or clear judgment and informed consent in the opinion of the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with All-cause mortality and Serious Adverse Events (SAEAs) | 6 months
  Investigational device safety with the intended study population with respect to 6 months follow up will be demonstrated using the following:
  All-cause mortality and Serious Adverse Events (SAEAs) throughout 6 months post-surgery.
Incidence of in-hospital procedure success. | up ot 24 hour.
  Success of the implant surgical procedure and ability to position the CORolla® TAA will be determined according to Implantation Rating Questionnaire.

SECONDARY OUTCOMES:
Rate of HF death and re-hospitalization due to HF (including IV diuretic) | 6 months
Rate of HF death and re-hospitalization due to HF (including IV diuretic) | 12 months
Rate, type and severity of procedure related and device-related events | 30 days
Rate of device related Major Adverse Cardiac and Neurological Events (MACNE) | up to 6 months
Change in Quality of Life (QoL) Questionnaire | up to 24 months
  Minnesota Living with Heart Failure.
Change in New York Heart Association functional Class (NYHA f. Cl). | up to 24 months
Change in exercise capacity as measured by the Six-Minute Walk test. | up to 24 months
Device impact on diastolic dysfunction markers assessed by conventional echocardiography imaging and novel approach including Tissue Doppler Imaging (TDI). | up to 24 months
  Composite measure: Left atrial volume index [ml/m^2], Early mitral flow velocity E [ml/sec], Mitral flow velocity during atrial systole A [ml/sec], E/A ratio, Mitral annular velocity e' [mm/sec], Declaration time [msec], E/e' [ml/mm], Left ventricular mass [gr], Ejection fiction [%], Pulmonary venous flow [m/sec], Transmitral flow propagation velocity [cm/sec].
Change of Wedge pressure | up to 24 months
  For safety assessment and impact of CORolla ® TAA therapy on this marker of diastolic dysfunction.
Change in Pulmonary Capillary Wedge Pressure during handgrip/ergometry | up to 24 months
  Applicable only to patients who are in a clinical condition that enables them to have the test and at sites that have the experience and the capabilities to perform this test.
Change in exercise testing during echocardiography | up to 24 months
  Composite measure: Maximal exercise tolerance defined as the number of metabolic equivalent (METs) at baseline and maximal: Early mitral flow velocity E [ml/sec], Mitral annular velocity e' [mm/sec] and E/e' [ml/mm]. Applicable only to patients who are in a clinical condition that enables them to have the test and at sites that have the experience to perform this test.
Change in VO2 Max | up to 24 months
  Applicable only to patients who are in a clinical condition that enables them to have the test and at sites that have the experience and the capabilities to perform this test.
Changes in cardiac medications, including daily diuretic dose. | up to 24 months
  The dose of furosemide [mg/d] and thiazide [mg/d] before and after the procedure and during follow up will be recorded and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- RAMBAM - Health Care Campus, Haifa, Israel

REFERENCES:
- See also: Company's website — http://www.corassist.com/